CLINICAL TRIAL: NCT06203470
Title: Efficacy and Safety of Mesobotox as a Potential New Therapeutic Modality of Psoriasis Vulgaris in Comparison/Combination With Topical Calcineurin Inhibitor
Brief Title: Botox Versus Tacrolimus in Psoriasis Vulgaris
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, SNIsrael, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTP
Record Dates: First submitted 2023-12-15; First posted 2024-01-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Botulinum Toxins, Type A; Tacrolimus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Botox group (Experimental): Patients will receive a single intradermal injection of Mesobotox as a monotherapy.
  Botulinum toxin injection: Botox injections will be intradermal. Concentration will be 100 U to be diluted with 5-ml sterile physiological sodium chloride solution. Each patient will receive individual injections of 1 U using a grid with points set at a distance of 1 cm apart. Up to two plaques per patient will be selected, whose diameter would not exceed 5-10 cm2. Each patient will receive a single BoNT-A injection
  Interventions: Drug: Botulinum Toxin-A
- Botox and Tacrolimus group (Experimental): Patients will receive a single intradermal injection of Mesobotox of the same dilution followed by topical application of Tacrolimus 0.03% ointment twice daily for 3 months.
  Interventions: Drug: Botulinum Toxin-A; Drug: Tacrolimus
- Tacrolimus group (Experimental): Patients will apply Tacrolimus (0.03%) as a monotherapeutic twice daily for 3 months
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Botulinum Toxin-A — Botulinum Toxin-A (BoNT-A) is an injectable neuromodulator produced by Clostridium Botulinum, a Gram-positive bacillus that causes Botulism.
  Arms: Botox and Tacrolimus group; Botox group
Drug: Tacrolimus — topical Calcineurin inhibitor
  Arms: Botox and Tacrolimus group; Tacrolimus group

SUMMARY:
Psoriasis is a systemic chronic relapsing immune-mediated disease which often requires a long-term therapy. Psoriasis occurs in around 2-3% of the total global population. In Egypt, the prevalence of psoriasis ranges between 0.19% and 3%.

Besides, it could have profound implications on the patients' psychological state and quality of life.

It is presented by erythematous, scaly plaques over the preferred sites. The pathogenesis of this highly complex disease is still far from being fully understood. Keratinocytes' hyperproliferation and immune system dysfunctions are well recognized contributors, with numerous treatments targeting these unique immunologic dysfunctions.

DETAILED DESCRIPTION:
Neurogenic inflammation has been suggested as an etiopathogenic factor of psoriasis. Previous reports revealed an increased concentration of nerve fibers as well as a high level of neuropeptides of cutaneous sensory nerve origin, primarily Substance P and calcitonin gene-related peptide (CGRP).

Some investigators reported improvement of psoriatic plaques after injuries that compromised peripheral nerves. Hence, it was postulated that cutaneous sensory afferent neurons are involved in the etiopathogenesis of psoriasis and may serve as a potential therapeutic target.

Substance P (SP) is a neuropeptide of sensory nerve origin that can influence the immune cell functions and the inflammatory responses in psoriasis. By binding to NK1R on T cells, SP can stimulate Th17 cell differentiation and production of interleukin-17A cytokine (IL-17A). IL-17A is a key effector cytokine in psoriasis, by releasing several pro-inflammatory cytokines, such as TNF alpha, stimulating abnormal keratinocytes' proliferation and promoting angiogenesis.

Topical drug therapy is the cornerstone of the treatment of mild to moderate psoriasis. It offers a direct skin targeting and avoids systemic adverse events. Several topical therapies are currently available for the treatment of psoriasis such as topical steroids, topical vitamin D3 analogues e.g. Calcipotriol, tar, anthraline, topical calcineurin inhibitors and tazarotene.

Tacrolimus, formerly known as FK506, is a macrolide antibiotic possessing immunosuppressive properties. Tacrolimus disrupts the intracellular activation of T-lymphocytes and inhibits the ability of calcineurin to regulate gene transcription. Thus, tacrolimus intervenes at an early stage of T-cell activation, leads to several secondary consequences providing effective and therapeutically efficient results to overcome problems associated with psoriatic skin disease.

Botulinum Toxin-A (BoNT-A) is an injectable neuromodulator produced by Clostridium Botulinum, a Gram-positive bacillus that causes Botulism. The clinical utility of BoNT-A originates from the ability to block muscular contractions by inhibiting neurotransmission between peripheral nerve cells and muscle fibers. Currently, BoNT-A is widely used for multiple aesthetic concerns that can be alleviated by local muscle relaxation, such as upper facial dynamic rhytides .

Botulinum Toxin-A can inhibit the release of neurotransmitters e.g. SP from the sensory motor neurons. SP is an important neuropeptide in the pathophysiological process of cutaneous neurogenic inflammation. Thus, it was hypothesized that BoNT-A can potentially be used for treating several inflammatory skin diseases, including psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of mild to moderate psoriasis vulgaris
* Patients who stopped any systemic therapy or phototherapy for at least 3 months and topical therapy for at least 4 weeks prior to enrollment.

Exclusion Criteria:

* • Psoriasis vulgaris involving > 10% of the body surface area, pustular or erythrodermic psoriasis.

  * Patients with neuromuscular disease or history of epilepsy.
  * Pregnant or lactating females.
  * Patients with any current dermatological disease.
  * Patients with any current systemic disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of Mesobotox for treatment of plaque psoriasis as a monotherapy versus its combination with a topical Calcineurin inhibitor 0.03% ointment and topical Calcineurin inhibitor 0.03% ointment alone. | 6 months
  This will be evaluated by measuring the (Psoriasis severity (TES) score) which is a physician-based, four-point scoring system in which the thickness, erythema, and scales within each plaque will be rated from 0 (none) to 3 (severe) to evaluate the therapeutic outcome within different groups before and after treatment.

SECONDARY OUTCOMES:
To explore the treatment effects on the histopathological features of psoriasis. | 2 months
  Three millimeter-punch biopsy specimens will be obtained before treatment, under local anesthesia from each patient and after 2 months of treatment. The biopsy specimens will be preserved in 10% formalin solution. Histopathological evaluation of treatment response will be performed using Hematoxylin and Eosin (H&E) stain.
To explore the treatment effects on the immunohistochemical features of psoriasis. | 2 months
  Immunohistochemical evaluation will be done using a special stain to detect SP before and 2 months after tratment.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Armstrong AW, Mehta MD, Schupp CW, Gondo GC, Bell SJ, Griffiths CEM. Psoriasis Prevalence in Adults in the United States. JAMA Dermatol. 2021 Aug 1;157(8):940-946. doi: 10.1001/jamadermatol.2021.2007. PMID 34190957
- [Background] Omar SS, Helaly HA. Prevalence of ocular findings in a sample of Egyptian patients with psoriasis. Indian J Dermatol Venereol Leprol. 2018 Jan-Feb;84(1):34-38. doi: 10.4103/ijdvl.IJDVL_1239_15. PMID 29067934
- [Background] Goff KL, Karimkhani C, Boyers LN, Weinstock MA, Lott JP, Hay RJ, Coffeng LE, Norton SA, Naldi L, Dunnick C, Armstrong AW, Dellavalle RP. The global burden of psoriatic skin disease. Br J Dermatol. 2015 Jun;172(6):1665-1668. doi: 10.1111/bjd.13715. Epub 2015 May 6. No abstract available. PMID 25645671
- [Background] Khattab FM, Samir MA. Botulinum toxin type-A versus 5-fluorouracil in the treatment of plaque psoriasis: Comparative study. J Cosmet Dermatol. 2021 Oct;20(10):3128-3132. doi: 10.1111/jocd.14306. Epub 2021 Jul 14. PMID 34146460
- [Background] Kubanov AA, Katunina OR, Chikin VV. Expression of Neuropeptides, Neurotrophins, and Neurotransmitters in the Skin of Patients with Atopic Dermatitis and Psoriasis. Bull Exp Biol Med. 2015 Jul;159(3):318-22. doi: 10.1007/s10517-015-2951-4. Epub 2015 Jul 24. PMID 26201903
- [Background] Popescu MN, Beiu C, Iliescu MG, Mihai MM, Popa LG, Stanescu AMA, Berteanu M. Botulinum Toxin Use for Modulating Neuroimmune Cutaneous Activity in Psoriasis. Medicina (Kaunas). 2022 Jun 16;58(6):813. doi: 10.3390/medicina58060813. PMID 35744076
- [Background] Khattab FM. Evaluation of Botulinum Toxin A as an Optional Treatment for Atopic Dermatitis. J Clin Aesthet Dermatol. 2020 Jul;13(7):32-35. Epub 2020 Jul 1. PMID 32983334
- [Background] Gonzalez C, Franco M, Londono A, Valenzuela F. Breaking paradigms in the treatment of psoriasis: Use of botulinum toxin for the treatment of plaque psoriasis. Dermatol Ther. 2020 Nov;33(6):e14319. doi: 10.1111/dth.14319. Epub 2020 Oct 8. PMID 32949180
- [Background] Zhang Y, Zhang H, Jiang B, Yan S, Lu J. A promising therapeutic target for psoriasis: Neuropeptides in human skin. Int Immunopharmacol. 2020 Oct;87:106755. doi: 10.1016/j.intimp.2020.106755. Epub 2020 Jul 28. PMID 32736190
- [Background] Chen SQ, Chen XY, Cui YZ, Yan BX, Zhou Y, Wang ZY, Xu F, Huang YZ, Zheng YX, Man XY. Cutaneous nerve fibers participate in the progression of psoriasis by linking epidermal keratinocytes and immunocytes. Cell Mol Life Sci. 2022 Apr 30;79(5):267. doi: 10.1007/s00018-022-04299-x. PMID 35488965
- [Background] Amalia SN, Uchiyama A, Baral H, Inoue Y, Yamazaki S, Fujiwara C, Sekiguchi A, Yokoyama Y, Ogino S, Torii R, Hosoi M, Ishikawa O, Motegi SI. Suppression of neuropeptide by botulinum toxin improves imiquimod-induced psoriasis-like dermatitis via the regulation of neuroimmune system. J Dermatol Sci. 2021 Jan;101(1):58-68. doi: 10.1016/j.jdermsci.2020.11.003. Epub 2020 Nov 6. PMID 33176965
- [Background] Barros PO, Ferreira TB, Vieira MM, Almeida CR, Araujo-Lima CF, Silva-Filho RG, Hygino J, Andrade RM, Andrade AF, Bento CA. Substance P enhances Th17 phenotype in individuals with generalized anxiety disorder: an event resistant to glucocorticoid inhibition. J Clin Immunol. 2011 Feb;31(1):51-9. doi: 10.1007/s10875-010-9466-6. Epub 2010 Sep 24. PMID 20865305
- [Background] Bera MM, Lu B, Martin TR, Cui S, Rhein LM, Gerard C, Gerard NP. Th17 cytokines are critical for respiratory syncytial virus-associated airway hyperreponsiveness through regulation by complement C3a and tachykinins. J Immunol. 2011 Oct 15;187(8):4245-55. doi: 10.4049/jimmunol.1101789. Epub 2011 Sep 14. PMID 21918196
- [Background] Wollina U, Tirant M, Vojvodic A, Lotti T. Treatment of Psoriasis: Novel Approaches to Topical Delivery. Open Access Maced J Med Sci. 2019 Aug 30;7(18):3018-3025. doi: 10.3889/oamjms.2019.414. eCollection 2019 Sep 30. PMID 31850114
- [Background] Kattimani V, Tiwari RVC, Gufran K, Wasan B, Shilpa PH, Khader AA. Botulinum Toxin Application in Facial Esthetics and Recent Treatment Indications (2013-2018). J Int Soc Prev Community Dent. 2019 Mar-Apr;9(2):99-105. doi: 10.4103/jispcd.JISPCD_430_18. Epub 2019 Apr 12. PMID 31058058
- [Background] Ward NL, Kavlick KD, Diaconu D, Dawes SM, Michaels KA, Gilbert E. Botulinum neurotoxin A decreases infiltrating cutaneous lymphocytes and improves acanthosis in the KC-Tie2 mouse model. J Invest Dermatol. 2012 Jul;132(7):1927-30. doi: 10.1038/jid.2012.60. Epub 2012 Mar 15. No abstract available. PMID 22418873
- [Background] Wallin EF, Hill DL, Linterman MA, Wood KJ. The Calcineurin Inhibitor Tacrolimus Specifically Suppresses Human T Follicular Helper Cells. Front Immunol. 2018 May 31;9:1184. doi: 10.3389/fimmu.2018.01184. eCollection 2018. PMID 29904381